CLINICAL TRIAL: NCT02912559
Title: Randomized Trial of Standard Chemotherapy Alone or Combined With Atezolizumab as Adjuvant Therapy for Patients With Stage III Colon Cancer and Deficient DNA Mismatch Repair
Brief Title: Combination Chemotherapy With or Without Atezolizumab in Treating Patients With Stage III Colon Cancer and Deficient DNA Mismatch Repair
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01417; NCI-2016-01417 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A021502 (Other: Alliance for Clinical Trials in Oncology); A021502 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2016-09-22; First posted 2016-09-23 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Colon Adenocarcinoma; DNA Repair Disorder; Lynch Syndrome; Stage III Colon Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; DNA Repair-Deficiency Disorders; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — atezolizumab; Specimen Handling; Fluorouracil; dehydroftorafur; Leucovorin; Magnetic Resonance Spectroscopy; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (combination chemotherapy, atezolizumab) (Experimental): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV as a bolus on day 1, then continuously over 46 hours on days 1-3 of each cycle. Treatment repeats every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive atezolizumab IV over 30-60 minutes on day 1 of each cycle, beginning in cycle 1 or 2. Treatment repeats every 14 days for up to 25 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI every 6 months for the first 2 years, then for years 3-5 or until evidence of relapse, whichever comes first. Patients may also undergo blood sample collection throughout the trial.
  Interventions: Drug: Atezolizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Other: Quality-of-Life Assessment
- Arm II (combination chemotherapy) (Active Comparator): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV as a bolus on day 1, then continuously over 46 hours on days 1-3 of each cycle. Treatment repeats every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI every 6 months for the first 2 years, then for years 3-5 or until evidence of relapse, whichever comes first. Patients may also undergo blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Leucovorin Calcium; Procedure: Magnetic Resonance Imaging; Drug: Oxaliplatin; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm I (combination chemotherapy, atezolizumab)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; Elplat; JM 83; JM-83; JM83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; RP54780; SR 96669; SR-96669; SR96669
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase III trial studies combination chemotherapy and atezolizumab to see how well it works compared with combination chemotherapy alone in treating patients with stage III colon cancer and deficient deoxyribonucleic acid (DNA) mismatch repair. Drugs used in combination chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving combination chemotherapy with atezolizumab may work better than combination chemotherapy alone in treating patients with colon cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether atezolizumab combined with fluorouracil (FOLFOX) and its continuation as monotherapy can significantly improve disease-free survival (DFS) compared to FOLFOX alone in patients with stage III colon cancers and deficient DNA mismatch repair (dMMR).

SECONDARY OBJECTIVES:

I. To determine whether atezolizumab combined with FOLFOX and its continuation as monotherapy can significantly improve overall survival compared to FOLFOX alone in patients with stage III colon cancers and dMMR.

II. To assess the adverse events (AE) profile and safety of each treatment arm, using the Common Terminology Criteria for Adverse Events (CTCAE) and patient related outcomes (PRO)-CTCAE (among patients aged >= 18 years).

QUALITY OF LIFE OBJECTIVE:

I. To determine the impact of the addition of atezolizumab to FOLFOX on patient-reported neuropathy, health-related quality of life (QOL), and functional domains of health-related QOL.

II. To access the efficacy of atezolizumab adjusting for baseline QOL and fatigue measurements.

POTENTIAL CORRELATIVE SCIENCE OBJECTIVES:

I. To determine if the "immunoscore" can predict the efficacy of atezolizumab for disease-free survival among patients with stage III colon cancer.

II. To assess whether circulating immune cell populations can predict the efficacy of atezolizumab as adjuvant therapy for stage III colon cancer.

III. To explore the associations of genomic alterations identified in cell-free (cf)DNA with DFS in patients treated with FOLFOX with or without atezolizumab.

IV. To assess whether soluble markers of systemic inflammation in blood can predict the efficacy of atezolizumab as adjuvant therapy for stage III colon cancer.

V. To assess the relationship between baseline plasma 25(OH) D levels, change in 25(OH)D levels, and DFS and overall survival (OS) in patients with stage III colon cancer receiving FOLFOX +/- atezolizumab.

VI. To determine the ability of using fecal microbiota and their metabolic products to predict survival benefit from anti-PD-L1 antibody therapy in dMMR colon cancer patients.

VII. To determine if hypermutation or hyper-indel status is associated with response to atezolizumab.

VIII. To determine if unique messenger ribonucleic acid (mRNA) expression signatures are predictive of disease-free survival among patients receiving adjuvant chemotherapy for stage III colon cancer.

IX. To determine if the efficacy of atezolizumab differs among dMMR cancers due to germline MMR mutation (MLH1, MSH2, MSH6, PMS2) versus those with MLH1 hypermethylation and CIMP in patients with stage III colon cancer.

X. To identify overall mutational burden and number of putative tumor neoantigens in colon carcinoma specimens.

XI. To determine changes in growth patterns compared to baseline (relative to age-specific standards for height and weight). (Patients aged 12 to < 18 years to evaluate the impact of atezolizumab on growth and development patterns in this population) XII. To determine changes in development patterns compared to baseline (relative to onset of menarche [for females] and pubertal changes). (Patients aged 12 to < 18 years to evaluate the impact of atezolizumab on growth and development patterns in this population)

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive oxaliplatin intravenously (IV) over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV as a bolus on day 1, then continuously over 46 hours on days 1-3. Treatment repeats every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive atezolizumab IV over 30-60 minutes starting on day 1 of cycle 1 or 2. Treatment repeats every 14 days for up to 25 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) every 6 months for the first 2 years, then for years 3-5 or until evidence of relapse, whichever comes first. Patients may also undergo blood sample collection throughout the trial.

ARM II: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV as a bolus on day 1, then continuously over 46 hours on days 1-3. Treatment repeats every 14 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI every 6 months for the first 2 years, then for years 3-5 or until evidence of relapse, whichever comes first. Patients may also undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up for recurrence every 6 months for 2 years, then annually for 3 years. Patients are also followed up for survival every 6 months for up to 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage III colon adenocarcinoma (any T [Tx, T1, T2, T3, or T4], N1-2M0; includes N1C); tumors must be deemed to originate in the colon including tumors that extend into/involve the small bowel (e.g. those at the ileocecal valve)
* Presence of deficient (d) DNA mismatch repair (dMMR); MMR status must be assessed by immunohistochemistry (IHC) for MMR protein expression (MLH1, MSH2, MSH6, PMS2) where loss of one or more proteins indicates dMMR; dMMR may be determined either locally or by site-selected reference lab; Note: loss of MLH1 and PMS2 commonly occur together; formalin-fixed paraffin-embedded (FFPE) tumor tissue is required for subsequent retrospective central confirmation of dMMR status
* Patients with testing that did not show dMMR (loss of MMR protein) are not eligible to participate; patients whose tumors show MSI-H by PCR-based assay are not eligible to participate unless they also have MMR testing by IHC and are found to have dMMR (i.e. loss of one or more MMR proteins)
* Patients who are known to have Lynch syndrome, have been found to carry a specific germline mutation in an MMR gene (MLH1, MSH2, MSH6, PMS2), and have been shown to be dMMR by IHC are eligible to participate
* Tumors must have been completely resected; in patients with tumor adherent to adjacent structures, en bloc R0 resection must be documented in the operative report or otherwise confirmed by the surgeon; near or positive radial margins are acceptable so long as en bloc resection was performed; proximal or distal margin positivity is not permitted
* Entire tumor must be in the colon (rectal involvement is an exclusion); surgeon confirmation that entire tumor was located in the colon is required only in cases where it is important to establish if the tumor is a colon versus (vs.) rectal primary; patients with more than one primary colon adenocarcinoma are eligible if the qualifying stage III tumor is confined to the colon, and not rectum, and the other cancers of lower stage are removed in the en bloc R0 resection
* Based upon the operative report and other source documentation, the location of the primary tumor will be categorized as proximal or distal to the splenic flexure (included with distal), and further categorization will be as follows: cecum/ascending, transverse, descending, sigmoid colon, or rectosigmoid colon
* No evidence of residual involved lymph node disease or metastatic disease at the time of registration based on clinician assessment of imaging; the treating physician will determine if incidental lesions on imaging require workup to exclude metastatic disease; if based on review of images, the treating physician determines the patient to be stage III, then the patient is eligible
* No prior medical therapy (chemotherapy, immunotherapy, biologic or targeted therapy) or radiation therapy for the current colon cancer except for one cycle of mFOLFOX6
* Age >= 12 years
* Performance Status:

  * Patients < 16 years of age: Lansky >= 50%
  * Patients 16 to < 18 years of age: Karnofsky >= 50%
  * Patients >= 18 years of age: Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* This study involves: 1) an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown; and 2) an agent that has known genotoxic, mutagenic, and teratogenic effects; therefore, for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required; a female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)
* Absolute neutrophil count (ANC) >= 1500 mm^3
* Platelet count >= 100,000 mm^3; platelets >= 75,000 required for patients who received cycle 1 of mFOLFOX6 prior to registration
* Creatinine =< 1.5 x upper limit of normal (ULN) or
* Calculated creatinine clearance >= 45 mL/min by Cockcroft-Gault equation

  * Alternatively, for patients < 18 years of age, maximum serum creatinine =< the below age-gender-specific norms:

    * 12 years: 1.2 (male and female)
    * 13 to < 16 years: 1.5 (male), 1.4 (female)
    * 16 to < 18 years: 1.7 (male), 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) except in the case of Gilbert disease
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Thyroid-stimulating hormone (TSH) within normal limits (WNL); supplementation is acceptable to achieve a TSH WNL; in patients with abnormal TSH, if free T4 is normal and patient is clinically euthyroid, patient is eligible
* No active known autoimmune disease, including colitis, inflammatory bowel disease (i.e. ulcerative colitis or Crohn's disease), rheumatoid arthritis, panhypopituitarism, adrenal insufficiency
* No known active hepatitis B or C

  * Active hepatitis B can be defined as:

    * Hepatitis B virus surface antigen (HBsAg) detectable for > 6 months;
    * Serum hepatitis B virus (HBV) DNA 20,000 IU/ml (105 copies/ml); lower values 2,000-20,000 IU/ml (104-105 copies/ml) are often seen in hepatitis B virus e antigen (HBeAg)-negative chronic hepatitis B
    * Persistent or intermittent elevation in ALT/AST levels
    * Liver biopsy showing chronic hepatitis with moderate or severe necroinflammation
  * Active hepatitis C can be defined as:

    * Hepatitis C antibody (AB) positive AND
    * Presence of hepatitis C virus (HCV) RNA
* Excluded if known active pulmonary disease with hypoxia defined as:

  * Oxygen saturation < 85% on room air, or
  * Oxygen saturation < 88% despite supplemental oxygen
* No grade >= 2 peripheral motor or sensory neuropathy
* Patients positive for human immunodeficiency virus (HIV) are eligible only if they meet all of the following:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL, and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests
* No other planned concurrent investigational agents or other tumor directed therapy (chemotherapy, radiation) while on study
* No systemic daily treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of registration
* No known history of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins
* No known hypersensitivity to Chinese hamster ovary (CHO) cell products or any component of the atezolizumab formulation
* No known allergy to 5-fluorouracil, oxaliplatin, or leucovorin

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | From the time from randomization to first documentation of disease recurrent or death, assessed up to 5 years
  DFS will be compared between treatment arms using the stratified log rank test at one-sided level 0.025. If zero DFS events are observed in a certain stratum at an interim analysis and unstratified log-rank is used, all subsequent analyses for DFS will use unstratified log-rank test. The hazard ratio (HR) for DFS will be estimated using a stratified Cox proportional hazards model and the 95 percent confidence interval (CI) for the HR will be provided. Results from an unstratified analysis will also be provided. Kaplan-Meier methodology will be used to estimate the median DFS for each treatment arm, and Kaplan-Meier curves will be produced. Brookmeyer Crowley methodology will be used to construct the 95 percent CI for the median DFS for each treatment arm.

SECONDARY OUTCOMES:
Overall survival | From the time from randomization to death, from any cause, assessed up to 5 years
  The distribution of overall survival will be estimated using the method of Kaplan-Meier. Overall survival will be compared between treatment arms using the log-rank test, only if DFS is statistically significant. The HR for OS will be estimated using a Cox proportional hazards model and the 95 percent CI for the HR will be provided. If a stratified log-rank test is used, stratified HR will be considered, and if an unstratified log-rank test is used, unstratified HR will be considered.
Incidence of adverse events | Up to 30 days after last treatment
  Assessed by Common Terminology Criteria for Adverse Events version 4.0. Frequency tables will be reviewed to determine the patterns. The overall adverse event rates will be compared between treatment arms using Chi-square test (or Fisher's exact test if the data in contingency table is sparse).

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Sinicrope, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (1052):
- United States (1029):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - John Muir Medical Center-Concord, Concord, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Ontario, Ontario, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - City of Hope West Covina, West Covina, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - AdventHealth Celebration, Celebration, Florida
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Phoebe Putney Memorial Hospital, Albany, Georgia
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta Oncology Associates PC-D'Antignac, Augusta, Georgia
  - Augusta Oncology Associates PC-Wheeler, Augusta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Freeport Memorial Hospital/Leonard C Ferguson Cancer Center, Freeport, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center, Moline, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - MercyOne Genesis Silvis Cancer Center, Silvis, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Baptist Health Floyd, New Albany, Indiana
  - Reid Health, Richmond, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - MercyOne Genesis Davenport Medical Center, Davenport, Iowa
  - MercyOne Genesis Davenport Cancer Center, Davenport, Iowa
  - Iowa Cancer Specialists, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Saint Elizabeth Healthcare Fort Thomas, Fort Thomas, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - Oncology Center of The South Incorporated, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Bloomfield, Bloomfield, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Michigan State University, East Lansing, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Covenant HealthCare Mackinaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Neurosurgeons of New Jersey-Ridgewood, Ridgewood, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - The Cancer Institute at Saint Francis Hospital, East Hills, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Cone Health Cancer Center at Asheboro, Asheboro, North Carolina
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Atrium Health Lincoln/LCI-Lincolnton, Lincolnton, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Trinity's Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Good Samaritan Hospital, Corvallis, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center in Greenville/UPMC Horizon, Greenville, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Cancer Center-Uniontown, Uniontown, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute at Pierre, Pierre, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Cookeville Regional Medical Center, Cookeville, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Thompson Cancer Survival Center - West, Knoxville, Tennessee
  - Thompson Oncology Group-Lenoir City, Lenoir City, Tennessee
  - Thompson Oncology Group-Maryville, Maryville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Thompson Oncology Group-Oak Ridge, Oak Ridge, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - Scott and White Healthcare Round Rock, Round Rock, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Ballad Health Cancer Care - Bristol, Bristol, Virginia
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Cancer Specialists of Tidewater Limited, Chesapeake, Virginia
  - Peninsula Cancer Institute-Gloucester, Gloucester, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Peninsula Cancer Institute-Newport News, Newport News, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Cancer Specialists of Tidewater-Suffolk, Suffolk, Virginia
  - Peninsula Cancer Institute-Cancer Specialists of Tidewater, Virginia Beach, Virginia
  - Peninsula Cancer Institute-Williamsburg, Williamsburg, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - FHCC at EvergreenHealth, Kirkland, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Germany (12):
  - Technical University Dresden, Dresden, Saxony
  - Charite Humboldt - University Hospital, Berlin
  - Saint Josef-Hospital Bochum, Bochum
  - Onkologie-Cologne, Cologne
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Hamatologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Universitaet Leipzig, Leipzig
  - Medizinische Universitat, Mannheim
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Medizinische Klinik Iii, München
  - University Hospital Ulm, Ulm
  - University Hospital Wuerzburg, Würzburg
- Puerto Rico (11):
  - Advance Oncology Center, Aguadilla
  - Doctor's Cancer Center-Arecibo, Arecibo
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Hematologia Oncologia San Pablo, Bayamón
  - HIMA San Pablo Oncologic Hospital, Caguas
  - Doctors Cancer Center, Manatí
  - Instituto Oncologia Moderna Ponce, Ponce
  - San Juan Community Oncology Group, San Juan
  - Primary Care Physician Group, San Juan
  - San Juan City Hospital, San Juan
  - Centro de Hematologia y Oncologia del Sur, Santa Isabel

REFERENCES:
- [Derived] Langenfeld SJ, Raman S, Gribovskaja-Rupp I. Selected Abstracts. Dis Colon Rectum. 2025 Oct 1;68(10):1224-1230. doi: 10.1097/DCR.0000000000003879. Epub 2025 Jul 9. No abstract available. PMID 40953502